CLINICAL TRIAL: NCT01898689
Title: Optimizing Local Anesthetic Concentration for Continuous Popliteal-Sciatic Nerve Blocks
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Professor of Anesthesiology, In Residence, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Baxter Popliteal Volunteer
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Results first posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Relatively Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: This is a split-body study in which each study subject receives both treatments: one on each side of the body. Which treatment is applied to which side of the body is randomized (and masked).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The only individual aware of the treatment group assignments is the investigational pharmacist who has no interaction with the study subjects. Treatment group assignments were released by the investigational pharmacy only after completion of data collection.
Oversight: Data Monitoring Committee: No

ARMS (2):
- RIGHT side Ropivacaine 0.1% and LEFT side Ropivacaine 0.4% (Experimental): Bilateral sciatic perineural catheters were inserted and ropivacaine administered as a basal infusion concurrently. For the right catheter, ropivacaine 0.1% was infused at 8 mL/h basal for 6 hours. For the left catheter, ropivacaine 0.4% was infused at 2 mL/h for 6 hours.
  Interventions: Drug: Ropivacaine 0.1%; Drug: Ropivacaine 0.4%
- RIGHT side Ropivacaine 0.4% and LEFT side Ropivacaine 0.1% (Active Comparator): Bilateral sciatic perineural catheters were inserted and ropivacaine administered as a basal infusion concurrently. For the right catheter, ropivacaine 0.4% was infused at 8 mL/h basal for 6 hours. For the left catheter, ropivacaine 0.1% was infused at 2 mL/h for 6 hours.
  Interventions: Drug: Ropivacaine 0.1%; Drug: Ropivacaine 0.4%

INTERVENTIONS:
Drug: Ropivacaine 0.1% — A sciatic catheter was inserted and ropivacaine 0.1% was administered as a basal infusion for 6 hours.
  Other Names: continuous peripheral nerve block
Drug: Ropivacaine 0.4% — A sciatic catheter was inserted and ropivacaine 0.4% was administered as a basal infusion for 6 hours.
  Other Names: continuous peripheral nerve block

SUMMARY:
A continuous peripheral nerve block-also termed "perineural local anesthetic infusion"-involves the insertion of a tiny tube (a "catheter") through the skin and adjacent to a peripheral nerve, followed by local anesthetic (numbing medicine) administration via the catheter, providing pain control following surgery. Continuous peripheral nerve blocks may be provided in the hospital setting, but the use of lightweight, portable pumps permits infusion at home as well. However, it remains unknown if the concentration of the local anesthetic influences the block effects; or, is it rather simply the total dose of medication that is important. If it is the latter, then the concentration of local anesthetic could be increased, allowing a decreased basal infusion rate, which would allow patients at home to receive twice the duration of potent pain control since their infusion pump local anesthetic reservoir would last twice as long as current practice. In addition, if one concentration/dose combination results in less muscle weakness, but with at least equivalent analgesia, then the risk of falling might be decreased as well.

The investigators will test the hypothesis that providing ropivacaine at different concentrations and rates (0.1% at 8 mL/hour vs. 0.4% at 2 mL/hour)-but at an equivalent total basal (8 mg/hour)-produces comparable effects when used in a continuous popliteal-sciatic nerve block.

DETAILED DESCRIPTION:
The investigators therefore propose a volunteer-based clinical trial testing the hypothesis that providing ropivacaine at different concentrations and rates (0.1% at 8 mL/hour vs. 0.4% at 2 mL/hour)-but at an equivalent total basal dose (8 mg/hour)-produces comparable effects when infused for a continuous popliteal-sciatic nerve block. The primary endpoint will be tolerance to cutaneous electrical current applied on the plantar aspect of the foot. This is an objective endpoint that has been validated in multiple previous publications and correlates with intra- and post-operative pain.

This investigation will be a randomized, observer-masked, controlled, split-body, human-subjects clinical trial.

Enrollment. Subjects will be volunteers of both sexes, age 18 and older. Volunteers will be solicited using newspaper advertisements, fliers, and an existing database of volunteers (IRB approved). If a volunteer meets inclusion/exclusion criteria and desires study participation, written, informed consent will be obtained. Selection for inclusion will not be based on race or socioeconomic status. The study population of interest includes men and women of all races and socioeconomic status. A urine pregnancy test will be administered to all women of childbearing age following written informed consent but before any study interventions. This urine test will be administered by CTRI nursing staff using standard, FDA-approved urine pregnancy testing devices.

Inclusion criteria for the trial will be: (1) age ≥ 18 years; and (2) willing to have bilateral femoral perineural catheters placed with a subsequent ropivacaine infusion and motor/sensory testing for 6 hours, requiring an overnight stay in the UCSD GCRC/CTRI to allow dissipation of local anesthetic infusion effects by the following morning. Exclusion criteria for the trial will be: (1) current daily analgesic use; (2) opioid use within the previous 4 weeks; (3) any neuro-muscular deficit of either femoral nerves and/or quadriceps muscles; (4) morbid obesity [weight > 35 kg/m2]; (5) pregnancy (as determined by a urine pregnancy test prior to any study interventions); and (6) incarceration. We expect to recruit a maximum of 30 healthy volunteers; with a target goal of 24 for the analysis. Selection for inclusion will not be based on gender, race, or socioeconomic status. The study population of interest includes men and women of all races and socioeconomic status. There will be no participants from vulnerable populations, such as pregnant women, children, or prisoners

Perineural catheter insertion. Following written, informed consent, subjects will be admitted to the UCSD CTRI and have demographic/morphometric data recorded (e.g., age, weight, height). An intravenous line will be placed in an upper extremity, followed by external monitors (pulse oximeter, blood pressure, and EKG), and oxygen by nasal cannula. Sedation will be provided with intravenous fentanyl (50 mcg) and/or midazolam (1 mg), or oral valium (10 mg) and/or dilaudid (4 mg), as necessary. Subjects will then have bilateral popliteal-sciatic perineural catheters placed using standard UC San Diego techniques as previously published by the current P.I.7,8

Treatment Group Assignment. Subjects will have the right-sided catheter randomly assigned to one of two treatment groups: a ropivacaine concentration of 0.1% or 0.4%. Subjects will act as their own controls, with the contralateral side receiving the alternative concentration. The Investigational Drug Service will prepare the randomization list as well as the two ropivacaine reservoirs and two electronic infusion pumps (SIGMA Spectrum Infusion System, Baxter Healthcare International, Deerfield, IL) used to infuse the ropivacaine. All pumps will be FDA approved for infusion of local anesthetic. The basal rate of each infusion will be determined by the ropivacaine concentration in each pump reservoir: 0.1% (8 mL/h) or 0.4% (2 mL/h). While the basal rate and bolus volume will differ for each concentration, the total dose of local anesthetic will be the same for both treatments (8 mg/h). The local anesthetic reservoirs will be contained within an opaque bag prepared by the Investigational Drug Service, and the infusion rates displayed on the pumps covered, ensuring masking for both the subjects and observers (clinical research nurse taking the measurements). Following 6 hours (48 mg), the infusions will be discontinued and the catheters removed.

Treatment Group Basal Rate (mL/h) Basal Dose (mg/h) Total Dose (mg in 6 h) Ropivacaine 0.1% 8 8 48 Ropivacaine 0.4% 2 8 48

The tubing from the pumps to the subjects will be gently wound at least 5 rotations and covered with opaque tape, masking which perineural catheter is receiving which treatment (ropivacaine is clear, so the flow through the clear tubing from the tape to the perineural catheters will not be visually distinguishable). Subjects will remain within the CTRI until the following morning at least until Hour 22 for the final measurement; or, until their perineural infusion sensory and motor effects have resolved. If a subject requests early withdrawal from the study, they will remain in the CTRI until their perineural infusion sensory and motor effects have resolved.

Outcome Measurements. The selected measures have established reliability and validity and minimal inter-rater discordance. Measurements will be performed at Hour 0 (baseline), and on the hour until Hour 14, as well as the following morning at Hour 22. In all cases, measurements will be taken in the supine position with the dominant side measured first, followed by the non-dominant side.

Tolerance of transcutaneous electrical stimulation: Sensory perception-depth of analgesia-will be evaluated using tolerance of transcutaneous electrical stimulation with the same quantitative procedure validated and used in multiple clinical trials. Electrocardiogram pads are placed on the lateral aspect of the plantar surface of the foot which is covered by the sciatic nerve distribution; and, the tolerance to cutaneous electrical current is obtained using a nerve stimulator. The current is increased from 0 mA until subjects detect the electrical current (up to a maximum of 80 mA), at which time the current is recorded and the nerve stimulator turned off.

Muscle strength: We will evaluate muscle strength with an isometric force electromechanical dynamometer to measure the force produced during a maximum voluntary isometric plantar-flexion (muscles innervated by the sciatic nerve). The dynamometer will be placed against the bed's foot board (immobile) and the subject will be asked to take 2 seconds to come to maximum effort contracting the target muscles, maintain this effort for 5 seconds, and then relax. The measurements immediately prior to perineural ropivacaine administration will be designated as baseline measurements, and all subsequent measurements will be expressed as a percentage of the pre-infusion baseline.

Food and Drink: Both food and accompanying beverages/water will be provided by the hospital and served by the nursing staff immediately following catheter insertion. Meals will be provided without charge to the study subjects. There is no restriction on oral intake following catheter insertion.

Statistical Analysis. Sample size calculations are based on the primary aim of determining the relationship between perineural ropivacaine concentration and continuous popliteal-sciatic nerve block effects. To this end, we will perform an equivalency trial with the primary endpoint designated as the maximum tolerance to transcutaneous electrical stimulation at Hour 6. We will aim to demonstrate that differing the concentration (0.1% vs. 0.4%) applied to different legs of each subject, but providing an equal total dose (8 mg/h) of ropivacaine through a popliteal-sciatic perineural catheter does not result in a significant difference in tolerance between legs at Hour 6. We will conclude that the interventions are equivalent if the 95% confidence interval for the mean difference in tolerance between legs is contained within the pre-specified tolerance interval of +/- 10 mA. This value is used as the minimally clinically-relevant current since it approximates the tolerated electrical current range at baseline of the general population-in other words, natural variability and therefore a relatively small amount of current to detect.4 Based on previously-published data,1,4 we assume the standard deviation of tolerance difference between legs is SD=13 mA. With n=24 subjects, we will correctly conclude equivalence with approximately 80% probability ("power"). Alternatively, if the population difference is 10 mA, we will correctly reject equivalence with probability 5%. The mean difference between treatments will be estimated by Analysis of Covariance (ANCOVA), using baseline tolerance difference as a covariate. Subjects will receive each of the two treatments applied randomly to the left and right legs.

The same analyses will be applied to the secondary endpoints. Profiles of the responses over time will be examined with spaghetti and mean plots. Further secondary analyses will include mixed-effects modeling of the repeated measures. These models account for the hierarchical correlation of paired measures from each subject over time, and will be used to test the effects of subject characteristics, including sex, height, weight, body mass index, and age. The model will also allow simultaneous analysis of all observations while accounting for within-subject correlation, which can improve the standard errors of the estimated differential at each time point. The within-subject correlation will be modeled via a subject-specific random intercept. This is similar to a compound symmetric correlation structure without a random effect. The change from baseline, Y, for subject i and time t will be modeled with the linear mixed-effect model:

Yi(t¬j) = Yi(0) β0 + 1{t¬j=1}β1 + … + 1{t¬j=9}β9 + bi + eij

where 1{t¬j=k} is 1 if t¬j=k and 0 otherwise. The subject-specific random intercepts bi and residuals eij are assumed to follow a Gaussian distribution. We will present the estimated difference at each hour with unadjusted p-values, and p-values adjusted using the single-step method for simultaneous inference from parametric models.

Analyses will be executed using R version 2.12 (http://www.r-project.org). Additional analyses will include the Mann-Whitney U for nonparametric comparisons and Fisher's exact test for categorical variables (InStat, GraphPad Software, San Diego, California, United States).

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 years
2. willing to have bilateral femoral perineural catheters placed with a subsequent ropivacaine infusion and motor/sensory testing for 6 hours, requiring an overnight stay in the UCSD GCRC/CTRI to allow dissipation of local anesthetic infusion effects by the following morning

Exclusion Criteria:

1. current daily analgesic use
2. opioid use within the previous 4 weeks
3. any neuro-muscular deficit of either femoral nerves and/or quadriceps muscles
4. morbid obesity [weight > 35 kg/m2]
5. pregnancy (as determined by a urine pregnancy test prior to any study interventions)
6. incarceration

We expect to recruit a maximum of 30 healthy volunteers; with a target goal of 24 for the analysis. Selection for inclusion will not be based on gender, race, or socioeconomic status. The study population of interest includes men and women of all races and socioeconomic status. There will be no participants from vulnerable populations, such as pregnant women, children, or prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-07; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, MD, MS, Principal Investigator — University California San Diego
Locations (1):
- University California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Madison SJ, Monahan AM, Agarwal RR, Furnish TJ, Mascha EJ, Xu Z, Donohue MC, Morgan AC, Ilfeld BM. A randomized, triple-masked, active-controlled investigation of the relative effects of dose, concentration, and infusion rate for continuous popliteal-sciatic nerve blocks in volunteers. Br J Anaesth. 2015 Jan;114(1):121-9. doi: 10.1093/bja/aeu333. Epub 2014 Sep 23. PMID 25248648

RESULTS

PARTICIPANT FLOW:
Groups:
- Right Side Ropivacaine 0.1%, Left Side Ropivacaine 0.4%: Ropivacaine 0.1% administered at 8 mL/h basal for 6 hours on the right side of the body while ropivacaine 0.4% administered at 2 mL/h basal for 6 hours on the left side of the body.
- Right Side Ropivacaine 0.4%, Left Side Ropivacaine 0.1%: Ropivacaine 0.4% administered at 2 mL/h basal for 6 hours on the right side of the body while ropivacaine 0.1% administered at 8 mL/h basal for 6 hours on the left side of the body.
Period: Overall Study
Arm/Group | Right Side Ropivacaine 0.1%, Left Side Ropivacaine 0.4% | Right Side Ropivacaine 0.4%, Left Side Ropivacaine 0.1%
Started | 10 | 14
Completed | 10 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Right Side: Ropivacaine 0.1%: Bilateral sciatic perineural catheters were inserted and ropivacaine infused as a basal infusion through both for 6 hours. The right side of the body received 0.1% at 8 mL/h and the left side of the body received 0.4% at 2 mL/h.
- Right Side: Ropivacaine 0.4%: Bilateral sciatic perineural catheters were inserted and ropivacaine infused as a basal infusion through both for 6 hours. The right side of the body received 0.4% at 2 mL/h and the left side of the body received 0.1% at 8 mL/h.
- Total: Total of all reporting groups
Arm/Group | Right Side: Ropivacaine 0.1% | Right Side: Ropivacaine 0.4% | Total
Number analyzed (Participants) | 10 | 14 | 24
Age, Categorical [Count of Participants; unit: Participants]
  Age: <=18 years | 0 | 0 | 0
  Age: Between 18 and 65 years | 10 | 14 | 24
  Age: >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 9
  Male | 8 | 7 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 14 | 24
Height [Mean (Standard Deviation); unit: cm] | 175 (11) | 175 (11) | 175 (11)
Weight [Mean (Standard Deviation); unit: kg] — Right side dominant
  kg | 87.0 (15.3) | 79.2 (16.1) | 81.0 (17.0)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.0 (3.6) | 26.3 (5.0) | 26.6 (4.4)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerance to Transcutaneous Electrical Stimulation
Description: Electrocardiogram pads are placed on the lateral aspect of the plantar surface of the foot which is covered by the sciatic nerve distribution; and, the tolerance to cutaneous electrical current is obtained using a nerve stimulator. The current is increased from 0 mA until subjects detect the electrical current (up to a maximum of 80 mA), at which time the current is recorded and the nerve stimulator turned off.
Time Frame: Hour 6
Population: Since this was a split-body study, we included each individual who received the treatment. Since each of the 24 subjects received each of the treatments, the overall number of participants analyzed was 24 for each of the treatments. For this reason, the Total number of subjects appears to be '48', when in fact it was 48 treated sides.
Measure: Mean (Standard Deviation); unit: mA (milliamperes)
Groups:
- Ropivacaine 0.1%: Bilateral sciatic perineural catheters are inserted and ropivacaine is infused as a basal infusion for 6 hours. The right side received 0.1% at 8 mL/h and the left side received 0.4% at 2 mL/h.
- Ropivacaine 0.4%: Bilateral sciatic perineural catheters are inserted and ropivacaine is infused as a basal infusion for 6 hours. The right side received 0.4% at 2 mL/h and the left side received 0.1% at 8 mL/h.
Arm/Group | Ropivacaine 0.1% | Ropivacaine 0.4%
Number analyzed (Participants) | 24 | 24
mA (milliamperes) | 27.0 (20.2) | 26.9 (20.4)
Statistical Analysis 1: Comparison: Ropivacaine 0.1% vs Ropivacaine 0.4%; The null and alternative hypotheses were thus: H0: m0.1%-m0.4% ≤ -10 or m0.1%-m0.4% ≥ 10 and Ha: -10 , m0.1%-m0.4% , 10 where m0.1% and m0.1% are the population means for tolerance to current under 0.1% and 0.4% ropivacaine, respectively. With 24 evaluable subjects, we had 90% power at the 0.05 significance level to detect equivalence of 0.1% and 0.4% ropivacaine concentration on the mean tolerance to transcutaneous electrical stimulation; Test type: Equivalence — The a priori equivalence region for the difference in means between the two concentrations was specified as +10 mA. This value was considered the minimal clinically relevant current since it approximates the tolerated electrical current range at baseline of the general population-in other words, natural variability and therefore a relatively small amount of current to detect; p = 0.02, Mixed Models Analysis — P-values from the TOST procedure were 0.02 and 0.03 for the mean being inside the lower and upper boundaries, respectively. (estimated mean difference of 0.2 mA; 90% CI 28.2 to 8.5); Mean Difference (Net) = 0.2, 90% CI 2-sided [-8.2 to 8.5]

2. Secondary Outcome: Maximum Tolerance to Transcutaneous Electrical Stimulation
Description: as for outcome 1
Time Frame: baseline, Hours 1-14 (except 6 which was the primary outcome) and Hour 22
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mA (milliamperes)
Groups:
- Ropivacaine 0.1%: Ropivacaine 0.1% administered at 8 mL/h basal for 6 hours on the right side of the body while ropivacaine 0.4% administered at 2 mL/h basal for 6 hours on the left side of the body.
- Ropivacaine 0.4%: Ropivacaine 0.4% administered at 2 mL/h basal for 6 hours on the right side of the body while ropivacaine 0.1% administered at 8 mL/h basal for 6 hours on the left side of the body.
Arm/Group | Ropivacaine 0.1% | Ropivacaine 0.4%
Number analyzed (Participants) | 24 | 24
mA (milliamperes)
  Baseline | 23 (2.5) | 22.5 (2.5)
  Hour 1 | 19 (1.5) | 20 (2.5)
  Hour 2 | 18 (1.2) | 19 (2.5)
  Hour 3 | 20 (2.5) | 20.4 (2.5)
  Hour 4 | 25 (3) | 21 (2)
  Hour 5 | 25 (2.5) | 24.5 (2.5)
  Hour 7 | 27 (2.5) | 26.5 (2.5)
  Hour 8 | 27 (2.5) | 27.5 (2.5)
  Hour 9 | 23 (2.5) | 23.5 (2.5)
  Hour 10 | 25 (2.5) | 24.5 (2.5)
  Hour 11 | 23.5 (2.5) | 24.3 (2.5)
  Hour 12 | 25 (2.5) | 22 (2)
  Hour 13 | 19.5 (1) | 21.2 (1)
  Hour 14 | 23.5 (2.5) | 21 (2)
  Hour 22 | 17 (1) | 17 (1)

3. Secondary Outcome: Percent of Maximum Voluntary Isometric Contraction Baseline (Quadriceps Femoris)
Description: Muscle strength was evaluated with an isometric force electromechanical dynamometer (MicroFET2, Lafayette Instrument Company, Lafayette, IN) to measure the force produced during a MVIC during plantar flexion. The dynamometer was placed against the bed's foot board (immobile) and the subjects asked to take 2 seconds to come to maximum effort plantar flexing, maintaining this effort for 5 seconds, and then relaxing. The measurements immediately prior to perineural ropivacaine administration were designated as baseline measurements, and all subsequent measurements expressed as a percentage of the pre-infusion baseline.
Time Frame: baseline, Hours 1-14 and Hour 22
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage change from baseline MVIC
Arm/Group | Ropivacaine 0.1% | Ropivacaine 0.4%
Number analyzed (Participants) | 24 | 24
percentage change from baseline MVIC
  Baseline | 100 (0) | 100 (0)
  Hour 1 | 90 (1.2) | 98 (1.5)
  Hour 2 | 8.1 (1.2) | 8.1 (1.2)
  Hour 3 | 81.5 (1.5) | 81.0 (1.5)
  Hour 4 | 71.0 (1.0) | 71.5 (1.0)
  Hour 5 | 66 (4.9) | 57 (1)
  Hour 6 | 57 (1.4) | 56 (1.4)
  Hour 7 | 58 (1) | 57 (1)
  Hour 8 | 61 (2.5) | 63 (2.5)
  Hour 9 | 67 (2.1) | 68 (2)
  Hour 10 | 68 (2) | 66 (2)
  Hour 11 | 70 (1.0) | 67 (1)
  Hour 12 | 72 (2.5) | 78.5 (2.5)
  Hour 13 | 80 (2.5) | 70 (2.5)
  Hour 14 | 78 (3) | 78 (3)
  Hour 22 | 96 (0.8) | 97 (1.1)

ADVERSE EVENTS:
Time Frame: 22 hours after baseline measurement
Groups:
- Ropivacaine 0.1%: Ropivacaine 0.1% at 8 mL/h basal for 6 hours
  perineural infusion: A continuous peripheral nerve block-also termed "perineural local anesthetic infusion"-involves the insertion of a tiny tube (a "catheter") through the skin and adjacent to a peripheral nerve, followed by local anesthetic (numbing medicine) administration via the catheter, providing pain control following surgery. Continuous peripheral nerve blocks may be provided in the hospital setting, but the use of lightweight, portable pumps permits infusion at home as well.
- Ropivacaine 0.4%: Ropivacaine 0.4% at 2 mL/h basal for 6 hours
  perineural infusion: A continuous peripheral nerve block-also termed "perineural local anesthetic infusion"-involves the insertion of a tiny tube (a "catheter") through the skin and adjacent to a peripheral nerve, followed by local anesthetic (numbing medicine) administration via the catheter, providing pain control following surgery. Continuous peripheral nerve blocks may be provided in the hospital setting, but the use of lightweight, portable pumps permits infusion at home as well.
Arm/Group | Ropivacaine 0.1% | Ropivacaine 0.4%
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No